CLINICAL TRIAL: NCT02876146
Title: Alveolar Echinococcosis: Parasite Viability and Innovative Markers for Follow-up of Patients Treated With Albendazole - EchinoVISTA Prospective Clinical Study
Brief Title: Alveolar Echinococcosis: Parasite Viability and Innovative Markers for the Follow-up of Patients Treated With Albendazole
Acronym: EchinoVISTA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: R/2011/41
Record Dates: First submitted 2016-08-16; First posted 2016-08-23 (Estimated); Last update posted 2021-08-23 (Actual); Status verified 2017-10

CONDITIONS: Alveolar Echinococcosis
Keywords: Albendazole; Benzimidazole; Echinococcus multilocularis; Alveolar echinococcosis; Liver Diseases
MeSH Terms: conditions — Alveolar echinococcosis; Echinococcosis; Liver Diseases | interventions — benzimidazole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Hepatic alveolar echinococcosis (Other): Follow-up of standardized clinical, biological, and imaging characteristics (according to the WHO-expert consensus). Albendazole treatment, 400 mg x 2/d (or mebendazole if adverse effects)
  Standardized earlier withdrawal of benzimidazole :
  * Patients with non operable hepatic AE lesion : Withdrawal of benzimidazole treatment for patients without metastasis or neighbouring lesions (PxN0M0) after at least 4 years when viability markers became negative (PET-CT, serological markers)
  * Curative hepatectomy : Earlier withdrawal of benzimidazole treatment for patients without metastasis or neighbouring lesions (PxN0M0) after one year (WHO guidelines : 2 years), if viability markers became negative. Close prospective follow-up after withdrawal (PET-CT, serological markers)
  Interventions: Drug: Benzimidazole

INTERVENTIONS:
Drug: Benzimidazole — Withdrawal of benzimidazole after 4 years (non operable AE) or one year after surgery (curative hepatectomy)
  Other Names: Standardized earlier withdrawal of albendazole

SUMMARY:
Study design to define improved management of patients with hepatic alveolar echinococcosis treated with albendazole and especially make appropriate and timely decision of treatment withdrawal .

Based on exploratory analysis of existing and newly developed biological and imaging exams, for diagnosis and follow-up, and study of the relationship of these markers to the viability of the parasite and/or the activity of the parasitic lesions The study included two series of patients: operated on (curative hepatectomy) // non-operated on

DETAILED DESCRIPTION:
Close follow-up of the patients, based on WHO guidelines (Brunetti, Acta tropica 2010), including albendazole bloods levels determination.

Clinical exam, sampling and storing (biobank) of blood specimens at inclusion, M1, M3, M6, M9, M12, M18, M24, M30, M36, M44, M48.

Additional sampling for operated on patients : M15 and M21.

Imaging each year (US, CT, PET-CT & RMI).

Preservation of operative specimens samples at -80°C: samples taken at different location (center and periphery of the lesions) and in distant non-infected liver, for further studies of the immune response, RNA detection, and albendazole dosages.

ELIGIBILITY:
Inclusion Criteria:

* hepatic alveolar echinococcosis
* without antiparasitic treatment or with antiparasitic treatment and hepatectomy programmed

Exclusion Criteria:

* Patients with exclusively extra-hepatic form of alveolar echinococcosis
* Women without effective contraception (Contraindication to benzimidazoles)
* The immunosuppressed patients or receiving an immunosuppressive treatment will not be the object of a stop of the post-operative treatment by albendazole on 1 year after the intervention of radical resection; they can be included in the study but will receive the albendazole during 2 years; this exclusion applies to the patients treated by liver transplant.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2012-06; Primary Completion 2021-08 (Actual); Study Completion 2021-08 (Actual)

PRIMARY OUTCOMES:
Ratio of non-operated on patients with negative viability markers after a 4 years benzimidazole treatment | 4 years after last inclusion

SECONDARY OUTCOMES:
Ratio of non-operated on patients without AE relapse after benzimidazole withdrawal | 7 years after last inclusion
  Benzimidazole withdrawal after 4 years, then 3 years of close follow-up
Ratio of operated on patients without AE relapse after benzimidazole withdrawal | 3 years after last inclusion
  Benzimidazole withdrawal one year after surgery, then 3 years of close follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric GRENOUILLET, PharmD, PhD, Study Chair — University Hospital Besançon; Carine RICHOU, MD, Principal Investigator — University Hospital Besançon

IPD SHARING:
Plan to Share IPD: No